CLINICAL TRIAL: NCT01701089
Title: An Open-Label, Parallel Group Study to Assess the Inhibition of Brain MAO-B by RO4602522 After Repeated Dosing in Patients With Alzheimer's Disease and in Healthy Control Subjects
Brief Title: A Study of RO4602522 in Patients With Alzheimer Disease and in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP28253
Record Dates: First submitted 2012-09-27; First posted 2012-10-04 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer, Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — sembragiline

ARMS (2):
- RO4602522 Group 1 (Experimental)
  Interventions: Drug: 11C-L-deprenyl-D2; Drug: RO4602522
- RO4602522 Group 2 (Experimental)
  Interventions: Drug: 11C-L-deprenyl-D2; Drug: RO4602522

INTERVENTIONS:
Drug: 11C-L-deprenyl-D2 — Intravenous injection of 11C-L-deprenyl-D2 before positron emission tomography (PET); up to 3 injections in total
Drug: RO4602522 — Multiple doses of RO4602522 for 14 days
  Arms: RO4602522 Group 1
Drug: RO4602522 — Multiple doses of RO4602522 for up to 17 days
  Arms: RO4602522 Group 2

SUMMARY:
This open-label, multiple dose, parallel group study will assess the monoamine oxidase in the brain by in vivo positron emission tomography (PET) and safety of RO4602522 in patients with Alzheimer disease and in healthy volunteers. Patients and volunteers will receive multiple doses of RO4602522 and up to three injections of C11-L-deprenyl-D2 used in the PET.

ELIGIBILITY:
Inclusion Criteria:

General:

* Adults between 50-80 years of age. Females must be of non-child-bearing potential or if of child-bearing potential must use an acceptable form of contraception
* Body mass index (BMI) 18.0-32.0 kg/m2 inclusive

Healthy volunteers:

* Healthy, with no clinically relevant finding on physical examination at screening and Day -1
* No suspicion of cognitive impairment/early dementia from neuropsychological battery as judged by the investigator
* Able to participate and willing to give informed consent, and comply with the study restrictions.

Alzheimer Disease (AD) patients:

* Probable Alzheimer's disease, based on the National Institute of Neurological and Communicative
* Disorders and Stroke (NINCDS/ADRDA) and DSM-IV criteria
* Have a MMSE score at screening between 17 and 26 inclusive
* Modified Hachinski Ischemia Scale score of </=4
* A neuroimaging evaluation of the brain by MRI which supports a diagnosis of AD, with no evidence of focal disease to account for dementia or MRI exclusion criteria
* Medications taken for symptomatic treatment of AD must be maintained on a stable dosage regimen for at least 1 month before Day 1.
* Able to participate in all scheduled evaluations
* The patient has an appropriate caregiver or community dwelling with caregiver capable of accompanying subject on all visits to the center as judged by the investigator.
* In the opinion of the investigator the patient and caregiver will be compliant and have a high probability of completing the study.
* Signed and dated written informed consent obtained from the patient, co-signed by the patient's closest relatives and legally authorized representative, as required by national law for patients that are incapable of giving informed consent.

Exclusion Criteria:

General:

* Any active disease of the gastrointestinal (GI) system, liver, or kidneys that could result in altered absorption, excess accumulation, or impaired metabolism or excretion of drugs, including a history of major upper or middle GI tract surgery or current significant chronic disease of the GI tract
* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the screening assessment
* History of cancer in the past five years, except for fully treated local basal carcinoma, or fully treated carcinoma in situ of cervix
* Any major illness occurring within 1 month prior to the screening examination or febrile illness within 5 days prior to first dose
* History of psychotropic medicine abuse
* At risk of suicide in the opinion of the investigator or having a Yes to question number 4 or 5 of the Suicidal Ideation section of the C-SSRS
* Administration of ionizing radiation or radioisotope for research, diagnostics test or therapy within 12 months prior to the present study which would exceed the local yearly radiation dose exposures for participation in research studies (except for dental x-rays, minimal plain films such as chest and ankle X-rays) or subjects who regularly work with ionizing radiation or radioactive material.
* Participation in a clinical study with an investigational drug within 3 months before screening
* Positive test for hepatitis B, hepatitis C, or HIV at screening
* Loss or donation of more than 450 mL blood in the 4 months before screening or donation of plasma within 14 days of screening.
* History of drug abuse or evidence of drug abuse in urine test performed at screening
* Current alcohol abuse, or regular intake of more than 2 units of alcohol daily
* Coffee (or tea) consumption > 5 cups per day or xanthine containing drinks >/1.5 liter/day

Healthy volunteers:

* Family history of Alzheimer's disease in 1st and 2nd degree relative under 75 years.
* Evidence or history of clinically significant neurological or psychiatric disorders.

AD Patients:

* Any neurological or psychiatric condition not specified in exceptions
* Previous immunization therapy for AD

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in monoamine oxidase (MAO-B) enzyme activity as measured by in vivo positron emission tomography (PET) | Days 1, 14, and between days 15 and 34
Pharmacokinetics: Plasma concentration of RO4602522 | Days 1, 8, 14, and between Days 15 and 34

SECONDARY OUTCOMES:
Reduction of 11C-L-deprenyl-D2 tracer uptake by in vivo positron emission tomography (PET) | Days 1, 14, and between days 15 and 34
Safety: incidence of adverse events | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Stockholm, Sweden